CLINICAL TRIAL: NCT03668041
Title: CSP #2016 - National Adaptive Trial for PTSD Related Insomnia
Brief Title: National Adaptive Trial for PTSD Related Insomnia
Acronym: NAP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Trazodone; Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Trazodone (Active Comparator): Participants who are assigned to take trazodone, an active study medication.
  Interventions: Drug: Trazodone
- Eszopiclone (Active Comparator): Participants who are assigned to take eszopiclone, an active study medication.
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator): Participants who are assigned to take a placebo, a non-active study medication.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Trazodone — Trazodone is approved by the Food and Drug Administration (FDA) for treating major depression in adults but not for PTSD. Although trazodone has not been approved by the FDA to treat insomnia or PTSD, some doctors have tried it for these purposes. The doses in this study will be lower than the doses used to treat depression.
  Arms: Trazodone
Drug: Eszopiclone — Eszopiclone is approved by the FDA for treating insomnia, but it's unknown if eszopiclone can help treat insomnia when it's related to PTSD. Some doctors have tried it for this purpose. The doses in this study will be the same as the doses used to treat insomnia. A small study found it to be helpful for treating patients with PTSD.
  Arms: Eszopiclone
Other: Placebo — The active study medications listed above will be compared with a placebo, which is a pill that looks like a study medication but has no medication in it.
  Arms: Placebo

SUMMARY:
Many Veterans with posttraumatic stress disorder (PTSD) have trouble sleeping or have frequent nightmares. So far, no medication has been approved for treatment of insomnia in PTSD. The purpose of this research study is to find out if taking medications called trazodone or eszopiclone can help decrease symptoms of insomnia in patients with PTSD. PTSD is a form of intense anxiety which sometimes results from severe trauma. Symptoms may include nightmares, flashbacks, troublesome memories, difficulty sleeping, poor concentration, irritability, anger, and emotional withdrawal. Insomnia is a disorder that can make it hard to fall sleep, stay asleep or cause a person to wake up too early and not be able to fall back to sleep.

DETAILED DESCRIPTION:
VA Cooperative Studies Program #2016 is a double-blind three-arm adaptive clinical trial to compare the efficacy of trazodone hydrochloride and eszopiclone to placebo, as adjunctive therapies in the treatment of insomnia symptoms among Veterans with military related PTSD, as measured by statistically significant difference in change from baseline in Insomnia Severity Index (ISI) total score at Week 12.

Participants will be male and female Veterans with PTSD and moderate levels of insomnia as measured on the ISI. Veterans who meet inclusion and exclusion criteria will be randomized within each site to receive trazodone hydrochloride, eszopiclone or placebo. Permuted blocks randomization will be used within each participating site. A mid-point interim analysis will be conducted wherein active treatment arms meeting early futility stopping criteria may be dropped. If all active treatment arms are dropped at the interim analysis, the study will be stopped at that time. Otherwise, the study will continue, and the remaining sample size will be allocated to the remaining study arms with equal randomization probabilities. Study drug dose will ideally be increased using a flexible dose titration schedule over the initial 3-week period, and the maximally tolerated dose will be continued until the week 12 assessment.

The Insomnia Severity Index (ISI) is the primary outcome measure for this study. The Clinician Administered PTSD Scale for DSM-V (CAPS-5) will be the key secondary outcome measuring change in PTSD symptoms. Other secondary outcomes that measure PTSD and sleep include the PTSD Checklist (PCL-5) and Pittsburgh Sleep Quality Index Scale-Addendum for PTSD (PSQI-A). Other secondary outcomes include brief questionnaire secondary measures of comorbid depression (PHQ-9), anxiety (GAD-7), quality of life (WHOQOL-BREF), treatment satisfaction questionnaire for medication (TSQM-9), smoking and alcohol consumption (Timeline Follow-Back, or TLFB), clinical global change (CGI-S), resource utilization (Service Utilization and Resources Form, or SURF). Safety measures include: Suicide Screening Questionnaire, review of Adverse events, and measuring anger and aggression (Dimension of Anger Reaction-5, or DAR-5).

This study is designed to serve as a well-powered "screen" for efficacious medications for the treatment of PTSD-related insomnia from among the medications already widely prescribed for this purpose within VA. Thus, this study is powered to detect differences between trazodone and eszopiclone versus placebo. The 3-arm design will require a sample size of 774 in the three arms (trazodone, eszopiclone and placebo), based on a drop out rate of 10%, to provide 85% probability to establish efficacy of the two active medications (trazodone and eszopiclone) when both have an effect size of 0.35 as compared to placebo.

VA bears a unique responsibility for addressing the limited efficacy of current evidence-based pharmacotherapy practices for PTSD. Since 2001, there have been only two FDA-approved medications for PTSD, both serotonin reuptake inhibiting antidepressants (SRIs), and SRIs have limited efficacy for military-related PTSD. This "efficacy gap" results in widespread polypharmacy for PTSD in VA, such that Veterans with antidepressant-resistant symptoms are treated, on average, with more than three psychotropic medications that present risks without clear benefit. In particular, SRI-resistant insomnia in military-related PTSD is a significant problem for VA, with 88% of these patients reporting clinically significant sleep impairment. In PTSD, sleep disturbances contribute importantly to impairments in quality of life, reduced social and vocational function, suicide risk, and poorer health. Effective treatment of persisting insomnia in PTSD is a sufficiently serious unmet need that the 2017 VA/DoD Clinical Practice Guideline for the Management of Posttraumatic Stress Disorder, called for "studies of non-benzodiazepine sedative/hypnotics." The purpose of the study is address this gap through testing the efficacy of three non-benzodiazepine hypnotics in comparison to placebo, representing the three medications or medication classes that are most commonly prescribed to Veterans with PTSD on an off-label basis and have yet to be tested in a definitive clinical trial. A novel aspect of this study is its implementation of an adaptive design in which arms would be dropped for evidence of futility based on pre-specified criteria at a designated interim analysis, intended to increase the efficiency of the trial and thereby improve the feasibility of its ambitious aim. The VA Cooperative Studies Program is uniquely suited to conduct this study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to comprehend and provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study (approximately 17 weeks from the date of being randomized)
3. Individuals, between the ages of 18 and 75 years
4. Allow digital recording of phone interviews
5. PTSD related to military service
6. Primary DSM-5 diagnosis of PTSD, assessed by structured interview using the CAPS-5
7. Total CAPS-5 score 23
8. ISI >15
9. Screening clinical laboratory tests without clinically significant abnormalities that would make study participation inappropriate, as determined by the site investigator with input, if needed, from the study chair
10. Electrocardiogram (ECG) at baseline without clinically significant abnormalities that would make study participation inappropriate, as determined by the site investigator with input, if needed, from the study chair and/or contingent upon approval by consulting medical physician.
11. Females of childbearing potential:

    1. Must have a negative pregnancy test during screening
    2. Must agree not to become pregnant or breastfeed during the course of the study
    3. Must be willing to use a reliable form of contraception for 16 weeks (during study treatment and for 2 weeks after taking the last dose) which includes: barrier contraceptives (male or female condoms with or without a spermicide, diaphragm or cervical cap with spermicide, or intrauterine device) and hormone-based therapy (contraceptive pills, intrauterine devices, or Depo-Provera®)
    4. Birth control for female participants is not necessary if surgically sterile or if with a partner with whom they are not capable of conceiving children (defined as a surgically sterile female by hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; surgically sterile male who has undergone a complete orchiectomy or successful vasectomy; or a same sex partner)
12. Agree to secure firearms while receiving study treatment
13. If individuals are undergoing evidence-based psychotherapy (EBT), which includes cognitive behavioral therapy (CBT), cognitive processing therapy (CPT), prolonged exposure therapy (PE), and/or stress inoculation therapy (SIT), they must have started these therapies at least 60 days prior to starting screening. If screening is started, and it is then discovered that EBT was started within 60 days prior to screening, participants must wait at least 60 days since staring the new EBT before they can complete the screening ISI, the screening PCL, and the Phone Assessment. (Supportive individual and group therapy is allowed)
14. Agreement to adhere to Lifestyle Considerations (see Section 5.3) throughout study participation
15. Clinical evidence of adequately treated sleep apnea or absence of sleep apnea having a severity that would make study participation problematic, established by meeting one of the criteria below:

    1. Clinical evidence of adequately treated sleep apnea with a continuous positive airway pressure (CPAP) or alternative treatment device (as defined in Section 8.1) (Participants can be reevaluated at least 30 days after screen failure.)
    2. If clinically tested, sleep study negative for sleep apnea or results indicating an Apnea-Hypopnea Index (AHI) < 23 within the past 6 months
    3. If tested for study eligibility, ApneaLink (or equivalent alternative device) result or other sleep study shows AHI < 23.

Exclusion Criteria:

1. Currently enrolled in any other interventional study unless prior approval is provided by the study team (It is a CSP policy that exemptions will be assessed for individual patients on a case-by-case basis. Exemptions require the agreement in writing of the following individuals or groups: (1) the SIs of both studies; (2) the Study Chairs of the involved studies; (3) the appropriate CSP Center Director(s); and (4) the VA Central IRB.)
2. Allergy and/or history of intolerance to trazodone hydrochloride and/or eszopiclone, or history of experiencing complex sleep behaviors (i.e., sleep walking, sleep driving, and/or engaging in other activities while not fully awake) while taking any sleep medication
3. A comorbid current or lifetime diagnosis of bipolar I disorder, bipolar II disorder, schizoaffective disorder, schizophrenia or delusional disorder, or current comorbid diagnosis of schizophreniform disorder, brief psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder or psychotic disorder not otherwise specified (NOS) according to Structured Clinical Interview for DSM-5 (SCID)-I-RV/P
4. History of moderate or severe traumatic brain injury (TBI) or history of gross structural damage as shown on MRI.
5. Positive urine test for an illicit substance, excluding cannabis, within the past 90 days prior to screening
6. Substance use meeting DSM-5 criteria for moderate or severe dependence (excluding nicotine) within the past 12 months prior to screening. (Note: Current mild dependence for alcohol and cannabis use is acceptable, but current mild dependence of any other substances is exclusionary.)
7. Inpatient psychiatric hospitalization within 30 days prior to screening
8. Suicidal or homicidal ideation with intent or plan to harm themselves or others within 90 days prior to screening
9. Chronic liver disease with two or more of the following occurring within the past six months: international normalized ratio (INR) greater than or equal to 1.7 (not on warfarin therapy), bilirubin greater than or equal to 2 mg/dL, serum albumin less than or equal to 3.5 g/dL, ascites, or encephalopathy (Participants can be reevaluated in 30 days)
10. Clinical and laboratory evidence of untreated hypothyroidism or hyperthyroidism
11. A corrected QT (QTc) interval greater than 470 ms
12. Unstable, serious medical condition or one requiring acute medical treatment, or planned hospitalization for extended care
13. Dementia, epilepsy, stroke, or current treatment with warfarin for anticoagulation
14. Taking any of the exclusionary medications listed in Appendix A. Note- an individual taking one of these medications for the sole purpose of improving sleep that elects to undergo an adequate wash-out period of at least 5 half-lives of the parent compound or active metabolite (e.g., for medications like diazepam), under the care of the individual's clinical provider, would not be excluded by this criterion.
15. Under criminal investigation or pending legal charges with potential incarceration
16. Individuals who lack stable contact information (including lack of a telephone number)
17. Participants who anticipate working during the hours of midnight to 6am during the course of study trial
18. Participants with narcolepsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Baseline to 12 weeks
  Change in the Insomnia Severity Index score from baseline to the 12-week follow-up will serve as the primary outcome. Possible range for ISI 0-28. Higher score indicates more severe insomnia problem(s).
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 | 12 weeks
  The scale consists of 20 DSM-5 symptoms rated on a 0-4 scale of how much that symptom bothered the individual in the prior month. Possible range for CAPS-5 total score 0-80, CAPS symptom cluster subscores of: Re-experiencing (B) 0-20, Avoidance (C) 0-8, Alteration in Cognition and Mood (D) 0-28, Hyperarousal (E) 0-24, Significant Distress (G) 0-12, and Dissociation (I) 0-8. Higher score indicates more severe PTSD.
Pittsburgh Sleep Quality Index Scale-Addendum for PTSD | 12 weeks
  It is a self-administered questionnaire that assesses sleep quality and disturbances over a 1-month period of time. The 7 items in the addendum generate a summary score, with three additional questions if memories or nightmares of a traumatic experience are present. Possible range for PSQI-A score 0-21, and possible range for each item 0-3. Higher PSQI-A score indicates worse quality of sleep.
Patient Health Questionnaire-9 | 12 weeks
  It is a tool to measure comorbid depression. This scale is frequently used in VA settings, has been well validated, and is a quick self-administered questionnaire. Possible range for PHQ-9 0-27. Higher score indicates more severe depression. 0-4: None/Minimal depression, 5-9: Mild depression, 10-14: Moderate depression, 15-19: Moderately severe depression, 20-27: Severe depression.
The World Health Organization Quality of Life | 12 weeks
  It is a 26-item self-administered questionnaire scaled to assess functioning and quality of life. Possible range for WHOQOL-BREF Overall 4-20, WHOQOL-BREF domain subscores of: Physical Health 4-20, Psychological 4-20, Social Relationships 4-20, and Environment 4-20. Higher score indicates better satisfaction with life.
Treatment Satisfaction Questionnaire for Medication-9 | 12 weeks
  It is a 9-item questionnaire to measure treatment satisfaction. TSQM-9 are scored on 3 domains: Effectiveness, Convenience, Global Satisfaction. Possible range for TSQM-9 domain scores 0-100. Higher score indicates higher satisfaction with medication.
Service Utilization and Resources Form | 12 weeks
  An abbreviated subset of the Service Utilization and Resources Form (SURF) assessment will be used to evaluate alcohol and other substance use (cannabis, smoking, and caffeine) using Timeline Follow-Back and resource utilization (e.g., outpatient medical and/or psychiatric visits and use of inpatient treatment and housing services). Questionnaire; no summary score.
PTSD Checklist | 12 weeks
  It is a brief questionnaire measure of PTSD symptom severity that is widely used within and outside VA. Possible range for PCL-5 0-80. Higher score indicates greater propensity for chronic and delayed PTSD.
Generalized Anxiety Disorder-7 Scale | 12 weeks
  It is a self-administered tool to assess anxiety. Possible range for GAD-7 0-21. Higher score indicates more severe anxiety disorder. 0-4: None/Minimal anxiety, 5-9: Mild Anxiety, 15-21: Severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: John H. Krystal, MD, Study Chair — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (35):
- United States (35):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - CERC (VISN1, West Haven, CT), West Haven, Connecticut
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Overton Brooks VA Medical Center, Shreveport, LA, Shreveport, Louisiana
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krystal JH, Chow B, Vessicchio J, Henrie AM, Neylan TC, Krystal AD, Marx BP, Xu K, Jindal RD, Davis LL, Schnurr PP, Stein MB, Thase ME, Ventura B, Huang GD, Shih MC; CSP 2016 Study Team. Design of the National Adaptive Trial for PTSD-related Insomnia (NAP Study), VA Cooperative Study Program (CSP) #2016. Contemp Clin Trials. 2021 Oct;109:106540. doi: 10.1016/j.cct.2021.106540. Epub 2021 Aug 18. PMID 34416369

DOCUMENTS (1):
  • Informed Consent Form (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT03668041/ICF_000.pdf